CLINICAL TRIAL: NCT06499402
Title: The Effect of Pregnant-controlled Sacral Massage on Mothers' Labor Pain, Perception, Process and Midwives' Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12345678
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Labor Pain; Labor
MeSH Terms: conditions — Labor Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- experimental group (Experimental)
  Interventions: Other: massage

INTERVENTIONS:
Other: massage — sacral massage
  Arms: experimental group

SUMMARY:
Our study aims to determine the effect of pregnant-controlled automatic sacral massage on mothers' labor pain, perception, process and midwives' satisfaction. The research was planned as a randomized controlled experimental study. A total of 112 women, 56 pregnant women in the experimental and control groups, will be included in the study. In this project, an automatic massage device will be used during the active phase (when the cervical opening is between 5-6 cm and 10 cm) and a massage device in line with the pregnancy-controlled sacral massage application protocol. Pregnant women are followed throughout the active phase of labor and indicators reflecting labor pain, progress of labor, and the health status of the mother and the baby are used with the "Individual Identification Form", "Visual Comparison Scale", "Labor Monitoring Form", "Mother's Birth Perception Scale (ADAS)". The satisfaction of midwives will be evaluated with the "Evaluation of Satisfaction Status of Midwives Form".

ELIGIBILITY:
Inclusion Criteria:

* Participating in the study voluntarily
* having a cervical dilatation of 5-6 cm,
* being between 38-40 weeks of pregnancy,- being a single fetus, having a cephalic presentation,
* having a fetal weight between 2.5-4 kg,
* having no vision-hearing problems,
* having communication and cooperation skills

Exclusion Criteria:

* having pregnancy complications
* Those who have acute inflammatory problems in soft tissues, skin or joints, burns, nerve injuries, open wounds, rheumatoid and gouty arthritis,
* those who have used any non-pharmacological methods will not be admitted.

Ages: 18 Days to 45 Days | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2024-08-22 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
stress | 1 day
  questionnaire, stress scale

SECONDARY OUTCOMES:
labor pain | 1 day
  pain scale, VAS